CLINICAL TRIAL: NCT06594900
Title: Muscle Growth and Development of Neuromuscular Capacities in Prepubertal Children - a Randomized Controlled Intervention Study
Brief Title: Development of Muscle Function in Prepubertal Children As a Response to Growth and Resistance Training
Acronym: decade-fit
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ralf Roth (Other)
Responsible Party: Sponsor-Investigator, Ralf Roth, Principal Investigator, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: decade-fit
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-09

CONDITIONS: Focus on Healthy Infants
Keywords: resistance training; strength training; children; prepubertal children; health; neuromuscular capacities; neurmuscular; development; crossfit; functional training; weigth training; neuromuscular adaptation; hormonal adaptation; structural adaptation; morphological adaptation; children development; physiological adaptation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): This group receives no training programme and just continues its life and physical activity as it used to do.
- Resistance training intervention (Experimental): The participants in the intervention group take part in a 20-week strength training programme in which they train twice a week for 60 min. The training programme focuses on strengthening the knee extensor muscles. Each training session consists of three phases: Warm-up, resistance training and coordination exercises.
  In the warm-up as well as coordination phase, full-body games are played to activate and challenge the children. The strength training phase forms the core of each session and includes exercises such as squats, lunges and step-ups. These exercises are performed in four sets of 8-12 repetitions, with the intensity being increased over time. The aim is to perform the exercises with great effort, but not to the point of complete exhaustion.
  Interventions: Behavioral: resistance training intervention

INTERVENTIONS:
Behavioral: resistance training intervention — The RT intervention focuses on knee extensor muscles, following current guidelines. Children will attend two supervised 1-hour sessions per week, proven sufficient for adaptations. Trained coaches and a scientific assistant, supported by master students, will document the sessions. Sessions are spaced 48 hours apart, totaling 40 over 20 weeks, with eight sessions between PRE and MID.
  Each session has three phases: warm-up, strength, and coordination. Warm-up involves whole-body games to increase heart rate and prepare for strength training. The strength phase, documented for effort and adjustments, includes squats, lunges, and step-ups, with intensity changes over time. Four sets of 8-12 repetitions per exercise are performed, aiming for strength increase and hypertrophy. Movements are done with great effort but not until voluntary failure.
  The coordination phase focuses on age-appropriate strength and motor skills through a circuit of challenges.
  Other Names: strength training; functional training; crossFit training
  Arms: Resistance training intervention

SUMMARY:
Healthy skeletal muscle development is crucial for a life-long quality of life. Childhood and puberty may be key periods for developing muscle growth and neuromuscular capacities, which are essential for bone-muscle interaction, metabolism, and participation in various sports. Even though the central role of physical activity in healthy physical development is well recognized, the decline in muscular fitness in today's children is alarming. This can lead to lasting deficits in muscle development and have a negative impact on overall health.

Well-designed resistance training (RT) could address this problem, since it has an effective positive impact on muscular strength, bone density, metabolism, and spontaneous physical activity especially in childhood. In general, muscles adapt according to physical activity stimuli. However, children show different responses to exercise and training. The physiologic differences, which are reflected in lower neuromuscular capacities and hormonal responses, but also in a better resistance to fatigue than in adults, are not yet fully understood. It is well established, that RT in children is safe, effective and has multiple benefits for health. However, the underlying mechanisms that lead to increased muscle strength are unclear and it is unknown how sustainable these are.

Today's common conception is that increased muscular strength is predominantly caused by neural adaptations and changes in muscle morphology due to lower androgenic responses are negligible.

Although higher neuromuscular adaptation potential is evident, it is still not sufficient to explain all strength increases, suggesting that additional mechanisms are involved in the process. Most studies are outdated, had methodological and statistical limitations, and many state-of-the-art methods have not yet been applied to children, hence, there is a need for a comprehensive, in-depth investigation to understand muscle adaptations to training and growth in children. With this better understanding of the impact and adaption to RT stimuli on neuromuscular and structural development the proposed project can serve as a foundation for more targeted prevention strategies.

The aim of this study is to investigate neuromuscular, hormonal, and morphological adaptations following 4 and 20 weeks of RT, while also examining their longitudinal retention through two consecutive follow-ups over 1.5 years. In this randomized controlled trial, state-of-the-art measurement methods are employed to accurately delve into mechanisms of adaptation, some of which have not yet used in children before due to limited time or infrastructure resources. The neuromuscular assessments include maximal and explosive strength of leg extensors, voluntary activation, motor unit decomposition, as well as central and peripheral neuromuscular fatigability. The hormonal changes are measured acutely (testosterone, cortisol, IGF-1 and growth hormone) and chronically (testosterone, progesterone and IGF-1) in response to one or several training sessions. Static and dynamic ultrasound imagining is used to quantify muscle size, fascicle shortening velocity and muscle architecture. This design allows in-depth insights into short- and long-term adaptations on several physiological levels to provide a novel mechanistic understanding of muscle growth and function in children.

The major innovation of this research is the integration of diverse scientific perspectives, combining insights from neuromuscular physiology, endocrinology, and muscle morphology to provide a holistic understanding of RT adaptations and development in children of both sexes.

This comprehensive approach can form the basis for future training programs, enabling next generations to better understand the potential impact of musculature on health.

ELIGIBILITY:
Inclusion Criteria:

* Able to travel 6 times to the Departement of Sports, Exercise and Health for the measurements
* Able to travel 2 times per week to CrossFit Basel GmbH for 20 weeks to participate on the training
* Able to verbally communicate pain or discomfort
* Signed informed consent information from the parents

Exclusion Criteria:

* Any acute or chronic medical condition
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.
* Regular participation in resistance training (incl. CrossFit®) in the previous year.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
maximal isometric voluntary contraction of knee extensor muscles | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Maximal isometric voluntary contraction (MVC) of knee extensor muscles refers to the level of maximal force, which can be transferred to a resisted dynamometer. It is highly adaptive from stimuli like training through mainly two pathway: by neuromuscular adaptation or muscle hypertrophy. Therefore, this is a sensitive measure during growth and resistance training intervention.
  The measurement of isometric MVC of knee extensor muscles will be performed in a seated position in a dynamometer (Isomed 2000, D. & R. Ferstl GmbH, Germany). The test subjects are fixed at a hip and knee angle of 120° and 60° respectively. According to Maffiuletti et al. (2016) the subjects are instructed to extend their legs as fast and forceful as possible and hold the contraction for 3-5s against lever arm of the dynamometer. After a familiarization attempt, the measurement is performed 2-5 times (until <5% difference between two trials) with a rest of 1 min in between. Peak torque will be used as outcome.

SECONDARY OUTCOMES:
Neuromuscular fatiguability | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Neuromuscular fatigue, the exercise-induced reduction of force generating capacity, is a complex phenomenon, which allows interesting insights into physiology.
  The neuromuscular fatigability protocol of knee extensor muscles consists of repeated 5s-MVCs with 5s of rest, in the same setup as the MVC-measurements. The procedure continues until the voluntary force fails to reach the target value of 60% of its initial MVC. The subjects are not informed of this criterion of task failure and only receive a child-friendly visual animation to ensure the timing and motivation, and strong verbal encouragement. To account for central and peripheral fatigue, magnetic nerve stimulations (as described above) are applied within the first, last and every 5th MVCs in between. The amplitude of the potentiated twitch torque is considered as indicator of peripheral fatigue. Determination of VA according to the section above will be analysed within every stimulation to account for central fatigue.
Power and explosive force | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Power is the product from force and speed and therefore another neuromuscular characteristic of the muscle. Explosive force is measured from the rate of torque development within the MVC measurements. The force of the first rise within 150ms is considered the rate of torque development.
  Power per body mass, determined from a vertical countermovement jump (CMJ), has been shown to be correlated to leg extension strength in children while representing a more natural movement. The CMJ will be performed on a force plate (Leonardo Mechanograph®, Novotec medical, Pforzheim, Germany) with arms akimbo. The instruction will be to jump as high as possible. After familiarization, each participant performs 2-5 trials, with the best of the two trials with &amp;amp;lt;5% difference being used for the analysis. The most important outcome parameter of this test is the maximum power output (peak power) normalized to body weight.
Voluntary activation | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Voluntary activation refers to the maximal percentage at which motor units can be synchronously activated during a contraction. The voluntary activation will be assessed using the interpolated twitch method. The most common method for this is electric nerve stimulation, which is associated with discomfort and pain, so that for the pediatric population the magnetic stimulation of the peripheral nerve is used, which has been validated against electrical stimulation and previously used in prepubertal children. Participants will be asked to perform 3-5 knee extension MVCs, in which doublet supramaximal stimulus (100% stimulator output) will be delivered to the femoral nerve to calculate the superimposed twitch (ST). Approximately three seconds after the end of the first MVC, a second supramaximal stimulus will be applied to determine the potentiated resting twitch (PT) to calculate voluntary activation according to the formula: (1 - (ST/PT)) x 100.
Muscle size | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Muscle size will be measured in vivo using B-mode ultrasonography (ACUSON Juniper, SIEMENS Healthineers, Erlangen, Germany). Vastus lateralis anatomical cross-sectional area will be measured in a prone position at 70 to 30% of muscle length with extended field of view ultrasonography using a 5.6 cm, 6.2-13.3 MHz, linear-array probe (12L3, Acuson 12L3). A trained operator gathers three high-quality ultrasound images per section. Muscle images will be then analysed using automated analysis software to reduce subjectivity. Furthermore, vastus lateralis volume will be calculated from the ACSA using the truncated cone formula, as well as PCSA from muscle volume and fiber length.
Motor unit activity | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Surface high-density electromyography (HD-EMG) can be used to determine the motor unit activity during voluntary contractions. HD-EMG will be recorded from the vastus lateralis during trapezoidal contractions at 25, 50 and 75% of MVC in the same position as previous MVCs. A lot of familiarizations and a child-friendly animation will ensure data quality of results. Prior to the recording, the skin will be shaved and cleaned using abrasive paste. The 64-channel equally spaced electrode matrix (GR08MM1305; OT Bioelettronica, Torino, Italy) will be placed on the determined muscle innervation zone in alignment with the muscle fiber orientation. In order to ensure identical placement of the electrode matrix at all the data collection points, its position will be painted on acetate sheets and photographed (as a backup method). Recruitment thresholds of distinct motor units, firing frequency spectrum and conduction velocity will be analyzed.
Acute and chronic hormonal changes | Resting concentrations: from enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each. Acute changes from one training session: in 2nd and 2nd-last week
  Sampling for analytical analysis will be performed using Dried Blood Spots (DBS) at the participants ear lobe from a drop of capillary blood. Resting concentrations to measure testosterone, IGF-1 and progesterone will be taken at the beginning of every laboratory measurement point. To assess acute changes of testosterone, GH, IGF-1 and cortisol following one session of RT, further samples will be taken from before and 15 min after the session according to the expected peak in those hormones45. These samples are taken in the second and second-last week of the training intervention at the same times of day in which the control group also takes part in an identical training session.
Muscle fascicle shortening velocity | From enrollment (PRE) to after 4 weeks of intervention (MID), to the end of Intervention (POST), as well as to the two Follow-ups after 9 month each.
  Muscle fascicle shortening velocity is a measure to describe muscle fiber properties and their changes through adaptation.
  Vastus lateralis muscle fascicle shortening velocity, amount of shortening and changes in pennation angle and muscle thickness will be assessed during the initial MVC employing two ultrasonography devices (ArtUS, Telemed, Mailand, Italy) and two 6 cm, 5.0-9.0 MHz, linear array probes (LF9-5N60-A3, ArtUS EXTH-1). Images will be captured during all three trials with a sampling rate higher than 60 frames per second. Both probes will be placed in line and parallel between the two aponeurosis of the vastus lateralis muscles and fixed using a custom-made cast to ensure minimal probe movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport, Exercise and Health, Basel, Basellandschaft, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided